CLINICAL TRIAL: NCT05139199
Title: Effectiveness of Auricular Point Acupressure in Improving Fatigue, Sleep Quality, Physical Activity and Quality of Life in Patients With Pancreatic Cancer Under Chemotherapy
Brief Title: Effectiveness of Auricular Point Acupressure in Improving Quality of Life in Patients With Pancreatic Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Taipei Veterans General Hospital, Taiwan (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2021-12-005A
Record Dates: First submitted 2021-07-29; First posted 2021-12-01 (Actual); Last update posted 2023-08-23 (Actual); Status verified 2022-08

CONDITIONS: Pancreatic Cancer
Keywords: Chemotherapy; Fatigue; Sleep Quality; Physical Activity; Quality of Life
MeSH Terms: conditions — Pancreatic Neoplasms; Fatigue; Sleep Initiation and Maintenance Disorders; Motor Activity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Auricular Point Acupressure (Experimental): A 1-month regimen of auricular point acupressure, comprising usual-care of approximately 15-20 point pressing each time,3 times a day, seven times peer week.
  Interventions: Behavioral: Auricular Point Acupressure group
- usual-care group (No Intervention): These participants follows the standard Chemotherapy follow-up consisting of counseling by nurses and doctors.

INTERVENTIONS:
Behavioral: Auricular Point Acupressure group — A 1-month regimen of auricular point acupressure, comprising usual-care of approximately 15-20 point pressing each time,3 times a day, seven times peer week.
  Arms: Auricular Point Acupressure

SUMMARY:
This study will investigate the effectiveness of auricular point acupressure in improving fatigue,sleep quality,physical activity and quality of life in patients with pancreatic cancer under chemotherapy in taiwan.

Hypothesis:

1. The fatigue in auricular point acupressure group is significant improving than usual-care group at 1st, 2nd, 3rd and 4th week.
2. The sleep quality in auricular point acupressure group is significant improving than usual-care group at 1st, 2nd, 3rd and 4th week.
3. The physical activity in auricular point acupressure group is significant improving than usual-care group at 1st, 2nd, 3rd and 4th week.
4. The quality of life in auricular point acupressure group is significant improving than usual-care group at 1st, 2nd, 3rd and 4th week.

DETAILED DESCRIPTION:
This study will investigate the effectiveness of auricular point acupressure in improving fatigue,sleep quality,physical activity and quality of life in patients with pancreatic cancer under chemotherapy in taiwan.

ELIGIBILITY:
Inclusion Criteria:

1. Paitent who aged over 20, with clear consciousness, is capable of communicating with Chinese, and is able to perform ear acupoints by himself/herself.
2. Pancreatic Cancer patients who received chemotherapy in inpatient and outpatient department.
3. The subject who agrees and is willing to participate in the research after explaining the purpose of the research.

Exclusion Criteria:

1. Patient who is younger than 20 years old, illiterate, or is unable to cooperate with intervention measures.
2. Patient who is not suitable for ear acupoint pressing after evaluated by the attending physician.

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2022-02-23 (Actual); Primary Completion 2023-08-01 (Actual); Study Completion 2023-08-01 (Actual)

PRIMARY OUTCOMES:
Quality of Life (EORTC QLQ-C30 ) | baseline
  This scale was evaluated by self-assessment of various clinical problems for a week.The EORTC QLQ-C30 consists three subscales with 30 questions.The EORTC QLQ-C30 included three subscales: functioning scales (15questions), symptom scales (13 questions), and global health status (2questions). The reliability and validity of Cronbach'α was 0.52-0.89. About the functional scale and the global health status, the higher the total score, the better the quality of life; the lower the score in the symptom scale, the better the quality of life.
Quality of Life (EORTC QLQ-C30 ) | 1st week after recruited
  This scale was evaluated by self-assessment of various clinical problems for a week.The EORTC QLQ-C30 consists three subscales with 30 questions.The EORTC QLQ-C30 included three subscales: functioning scales (15questions), symptom scales (13 questions), and global health status (2questions). The reliability and validity of Cronbach'α was 0.52-0.89. About the functional scale and the global health status, the higher the total score, the better the quality of life; the lower the score in the symptom scale, the better the quality of life.
Quality of Life (EORTC QLQ-C30 ) | 2nd week after recruited
  This scale was evaluated by self-assessment of various clinical problems for a week.The EORTC QLQ-C30 consists three subscales with 30 questions.The EORTC QLQ-C30 included three subscales: functioning scales (15questions), symptom scales (13 questions), and global health status (2questions). The reliability and validity of Cronbach'α was 0.52-0.89. About the functional scale and the global health status, the higher the total score, the better the quality of life; the lower the score in the symptom scale, the better the quality of life.
Quality of Life (EORTC QLQ-C30 ) | 3rd week after recruited
  This scale was evaluated by self-assessment of various clinical problems for a week.The EORTC QLQ-C30 consists three subscales with 30 questions.The EORTC QLQ-C30 included three subscales: functioning scales (15questions), symptom scales (13 questions), and global health status (2questions). The reliability and validity of Cronbach'α was 0.52-0.89. About the functional scale and the global health status, the higher the total score, the better the quality of life; the lower the score in the symptom scale, the better the quality of life.
Quality of Life (EORTC QLQ-C30 ) | 4th week after recruited
  This scale was evaluated by self-assessment of various clinical problems for a week.The EORTC QLQ-C30 consists three subscales with 30 questions.The EORTC QLQ-C30 included three subscales: functioning scales (15questions), symptom scales (13 questions), and global health status (2questions). The reliability and validity of Cronbach'α was 0.52-0.89. About the functional scale and the global health status, the higher the total score, the better the quality of life; the lower the score in the symptom scale, the better the quality of life.
Quality of Life (EORTC QLQ-PAN26 ) | baseline
  This scale was evaluated by self-assessment of various clinical problems for a week.The EORTC QLQ-PAN26 consists of two subscales with 26 questions.The EORTC QLQ-PAN26 included two subscales：functioning scales (4 questions),symptom scales (22 questions). The reliability and validity of Cronbach'α was 0.69-0.97. About the functional scale, the higher the total score, the better the quality of life; the lower the score in the symptom scale, the better the quality of life.
Quality of Life (EORTC QLQ-PAN26 ) | 1st week after recruited
  This scale was evaluated by self-assessment of various clinical problems for a week.The EORTC QLQ-PAN26 consists of two subscales with 26 questions.The EORTC QLQ-PAN26 included two subscales：functioning scales (4 questions),symptom scales (22 questions). The reliability and validity of Cronbach'α was 0.69-0.97. About the functional scale, the higher the total score, the better the quality of life; the lower the score in the symptom scale, the better the quality of life.
Quality of Life (EORTC QLQ-PAN26 ) | 2nd week after recruited
  This scale was evaluated by self-assessment of various clinical problems for a week.The EORTC QLQ-PAN26 consists of two subscales with 26 questions.The EORTC QLQ-PAN26 included two subscales：functioning scales (4 questions),symptom scales (22 questions). The reliability and validity of Cronbach'α was 0.69-0.97. About the functional scale, the higher the total score, the better the quality of life; the lower the score in the symptom scale, the better the quality of life.
Quality of Life (EORTC QLQ-PAN26 ) | 3rd week after recruited
  This scale was evaluated by self-assessment of various clinical problems for a week.The EORTC QLQ-PAN26 consists of two subscales with 26 questions.The EORTC QLQ-PAN26 included two subscales：functioning scales (4 questions),symptom scales (22 questions). The reliability and validity of Cronbach'α was 0.69-0.97. About the functional scale, the higher the total score, the better the quality of life; the lower the score in the symptom scale, the better the quality of life.
Quality of Life (EORTC QLQ-PAN26 ) | 4th week after recruited
  This scale was evaluated by self-assessment of various clinical problems for a week.The EORTC QLQ-PAN26 consists of two subscales with 26 questions.The EORTC QLQ-PAN26 included two subscales：functioning scales (4 questions),symptom scales (22 questions). The reliability and validity of Cronbach'α was 0.69-0.97. About the functional scale, the higher the total score, the better the quality of life; the lower the score in the symptom scale, the better the quality of life.

SECONDARY OUTCOMES:
Fatigue(Brief Fatigue Inventory-Taiwan , BFI-T) | baseline
  This scale was evaluated by self-assessment of various clinical problems for 24 hours.The BFI-T have 9 questions. Retest reliability was 0.89-0.91.
Fatigue(Brief Fatigue Inventory-Taiwan , BFI-T) | 1st week after recruited
  This scale was evaluated by self-assessment of various clinical problems for 24 hours.The BFI-T have 9 questions. Retest reliability was 0.89-0.91.
Fatigue(Brief Fatigue Inventory-Taiwan , BFI-T) | 2nd week after recruited
  This scale was evaluated by self-assessment of various clinical problems for 24 hours.The BFI-T have 9 questions. Retest reliability was 0.89-0.91.
Fatigue(Brief Fatigue Inventory-Taiwan , BFI-T) | 3rd week after recruited
  This scale was evaluated by self-assessment of various clinical problems for 24 hours.The BFI-T have 9 questions. Retest reliability was 0.89-0.91.
Fatigue(Brief Fatigue Inventory-Taiwan , BFI-T) | 4th week after recruited
  This scale was evaluated by self-assessment of various clinical problems for 24 hours.The BFI-T have 9 questions. Retest reliability was 0.89-0.91.
Sleep quality(Pittsburgh Sleep Quality Index ) | baseline
  The Pittsburgh Sleep Quality Index (PSQI) consists of 19 self-rated questions and 5 questions rated by the bed partner or roommate. The reliability and validity of Cronbach'α was 0.83. About lower scores the higher the total score, the better the quality of sleep.
Sleep quality(Pittsburgh Sleep Quality Index ) | 1st week after recruited
  The Pittsburgh Sleep Quality Index (PSQI) consists of 19 self-rated questions and 5 questions rated by the bed partner or roommate. The reliability and validity of Cronbach'α was 0.83. About lower scores the higher the total score, the better the quality of sleep.
Sleep quality(Pittsburgh Sleep Quality Index ) | 2nd week after recruited
  The Pittsburgh Sleep Quality Index (PSQI) consists of 19 self-rated questions and 5 questions rated by the bed partner or roommate. The reliability and validity of Cronbach'α was 0.83. About lower scores the higher the total score, the better the quality of sleep.
Sleep quality(Pittsburgh Sleep Quality Index ) | 3rd week after recruited
  The Pittsburgh Sleep Quality Index (PSQI) consists of 19 self-rated questions and 5 questions rated by the bed partner or roommate. The reliability and validity of Cronbach'α was 0.83. About lower scores the higher the total score, the better the quality of sleep.
Sleep quality(Pittsburgh Sleep Quality Index ) | 4th week after recruited
  The Pittsburgh Sleep Quality Index (PSQI) consists of 19 self-rated questions and 5 questions rated by the bed partner or roommate. The reliability and validity of Cronbach'α was 0.83. About lower scores the higher the total score, the better the quality of sleep.
Physical Activity(3-d Physical Record;Three-day activity record) | baseline
  The design to estimate energy expenditure. Two days could be any day of the week, but the 3rd day had to be either a Saturday or a Sunday. A day was divided into 96 periods of 15 mins each, energy expenditure was qualified on a scale from 1 to 9.
Physical Activity(3-d Physical Record;Three-day activity record) | 1st week after recruited
  The design to estimate energy expenditure. Two days could be any day of the week, but the 3rd day had to be either a Saturday or a Sunday. A day was divided into 96 periods of 15 mins each, energy expenditure was qualified on a scale from 1 to 9.
Physical Activity(3-d Physical Record;Three-day activity record) | 2nd week after recruited
  The design to estimate energy expenditure. Two days could be any day of the week, but the 3rd day had to be either a Saturday or a Sunday. A day was divided into 96 periods of 15 mins each, energy expenditure was qualified on a scale from 1 to 9.
Physical Activity(3-d Physical Record;Three-day activity record) | 3rd week after recruited
  The design to estimate energy expenditure. Two days could be any day of the week, but the 3rd day had to be either a Saturday or a Sunday. A day was divided into 96 periods of 15 mins each, energy expenditure was qualified on a scale from 1 to 9.
Physical Activity(3-d Physical Record;Three-day activity record) | 4th week after recruited
  The design to estimate energy expenditure. Two days could be any day of the week, but the 3rd day had to be either a Saturday or a Sunday. A day was divided into 96 periods of 15 mins each, energy expenditure was qualified on a scale from 1 to 9.
Physical Activity(Exercise Counseling and Programming Preferences) | baseline
  Exercise preferences were assessed by questions related to exercise counseling and exercise programming.

CONTACTS AND LOCATIONS:
Overall Officials: Hui-Mei Chen, PhD, Study Chair — National Taipei University of Nursing and Health Sciences
Locations (1):
- Taipei Veterans General Hospital, Taipei County, Taiwan

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in this article, after deidentification (text, tables, figures, and appendices)
Supporting Information: Study Protocol
Time Frame: Beginning 12 months and ending 36 months following article publication
Access Criteria: Researchers who provide a methodologically sound proposal and receive the authors consent.

REFERENCES:
- [Derived] Gao WL, Chen HM, Liu CY, Huang TH, Li CP, Hsu SJ, Lee PC, Lee KC. Effects of Auricular Acupressure on Fatigue, Sleep Quality, Physical Activity, and Quality of Life in Pancreatic Cancer Patients Undergoing Chemotherapy: A Randomized Controlled Trial. Cancer Nurs. 2025 Apr 18. doi: 10.1097/NCC.0000000000001498. Online ahead of print. PMID 40179142